CLINICAL TRIAL: NCT03203200
Title: A Cognitive Behavioral And Structural HIV Prevention Intervention for Young Ugandan Women Engaging in High Risk Sexual Behavior
Brief Title: A Cognitive Behavioral And Structural HIV Prevention Intervention for Young Ugandan Sex Workers
Acronym: ZETRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Connecticut (Other); MRC/UVRI and LSHTM Uganda Research Unit (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01 HD085805-01; 5R01MH109337-02 (NIH)
Record Dates: First submitted 2017-02-24; First posted 2017-06-29 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Sexually Transmitted Infection
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- health literacy and technology skill building (Experimental): ZETRA cognitive behavioral and structural
  Interventions: Behavioral: ZETRA cognitive behavioral structural
- Standard Counselling (No Intervention): Standard of care prevention counselling

INTERVENTIONS:
Behavioral: ZETRA cognitive behavioral structural — ZETRA cognitive behavioral structural
  Arms: health literacy and technology skill building

SUMMARY:
This study develops and tests a behavioural and structural intervention to prevent unprotected sex among young female sex workers. Half the participants will receive the intervention and half will receive the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* HIV-uninfected women, aged 15-24 years, being sexually active and having engaged in any form of transactional sex at least once in the last 3 months, agreeing to participate in all intervention sessions and to all study procedures and interviews planned over 18 months of follow-up.

Exclusion Criteria:

* presence of any physical or mental condition likely to cause inability to provide consent or hinder study participation; HIV infection

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 640 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Unprotected Sex | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Rachel King, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Uganda Virus Research Institute, Entebbe, Uganda

REFERENCES:
- [Derived] King R, Muhanguzi E, Nakitto M, Mirembe M, Kasujja FX, Bagiire D, Seeley J. Mobility study of young women who exchange sex for money or commodities using Google Maps and qualitative methods in Kampala, Uganda. BMJ Open. 2021 May 19;11(5):e043078. doi: 10.1136/bmjopen-2020-043078. PMID 34011583